CLINICAL TRIAL: NCT03309358
Title: A Multiple-Site, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose (SAD) Study to Assess the Safety and Tolerability of Inhaled SNSP113 in Healthy Male Subjects (Part A) and Subjects With Stable Cystic Fibrosis (Part B)
Brief Title: A Study of the Safety and Tolerability of Inhaled SNSP113 in Healthy Subjects and Subjects With Stable Cystic Fibrosis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Successful completion of Part A. Company decision to end early.
Sponsor: Synspira, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: SNSP113-17-101
Record Dates: First submitted 2017-10-05; First posted 2017-10-13 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Lung Diseases; Pulmonary Disease; Cystic Fibrosis; Cystic Fibrosis Lung; Cystic Fibrosis Pulmonary Exacerbation; Cystic Fibrosis With Exacerbation; Respiratory Tract Disease; Pulmonary Inflammation; Multi-antibiotic Resistance; Antibiotic Resistant Infection; Lung Infection; Lung Infection Pseudomonal; Lung; Infection, Atypical Mycobacterium; Burkholderia Infections; Burkholderia Cepacia Infection; Lung Inflammation
Keywords: Cystic Fibrosis; Pulmonary exacerbation; Pulmonary inflammation; Respiratory tract disease; Pulmonary disease; Biofilms
MeSH Terms: conditions — Lung Diseases; Cystic Fibrosis; Respiratory Tract Diseases; Pneumonia; Infections; Mycobacterium Infections, Nontuberculous; Burkholderia Infections

STUDY DESIGN:
Intervention Model Description: This is a multiple-site, randomized, double-blind, placebo-controlled, single ascending dose (SAD) study to assess the safety and tolerability of inhaled SNSP113 in healthy subjects (Part A) and subjects with stable CF (Part B).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inhaled SNSP113 (Experimental)
  Interventions: Drug: Inhaled SNSP113
- Inhaled Placebo (Placebo Comparator)
  Interventions: Drug: Inhaled Placebo

INTERVENTIONS:
Drug: Inhaled SNSP113 — A single ascending dose of inhaled SNSP113 will be administered to healthy subjects and subjects with stable cystic fibrosis.
  Arms: Inhaled SNSP113
Drug: Inhaled Placebo — A single dose of inhaled placebo control will be administered to healthy subjects and subjects with stable cystic fibrosis.
  Arms: Inhaled Placebo

SUMMARY:
Although Cystic Fibrosis is a complex genetic disease affecting many organs, lung disease is the primary cause of mortality. The objective of this study is to determine the safety and tolerability of SNSP113 in healthy subjects and subjects with stable cystic fibrosis.

ELIGIBILITY:
Inclusion Criteria:

Part A

* Healthy male adults ≥18 and ≤50 years of age at screening.
* Baseline FEV1 80-120% of predicted at Screening.
* Oxygen saturation of ≥ 96% on room air as determined by pulse oximetry at Screening.
* Screening laboratory tests within normal limits.

Part B

* Female and Male subjects who are ≥18 years of age and a confirmed diagnosis of CF.
* FEV1 >50% of predicted.
* Oxygen saturation of ≥ 94% on room air as determined by pulse oximetry at Screening.
* Stable CF pulmonary disease as judged by the Investigator.

Exclusion Criteria:

Part A

* Any history of any form of lung disease or any systemic disease that may affect the lung or pulmonary function.
* Former regular smoker or has smoked tobacco or cannabis products within the last 30 days.
* Any history of any form of liver disease, renal disease, cardiac disease, hematologic disease, neurologic disease, atopy or any chronic condition.
* Participation in one or more healthy subject studies within the prior 3 months.

Part B

* Participation in a clinical trial involving receipt of an investigational product within the 30 days prior to screening.
* Female subjects who are pregnant (a negative serum pregnancy test must be demonstrated at screening), have a positive pregnancy test, are lactating or who plan to become pregnant within 90 days after dosing.
* Subjects requiring supplemental oxygen.
* Hemoptysis of >5 mL within 12 weeks of screening.
* Listed for organ transplantation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy Male Subjects, Part A
  Female and Male Subjects with Stable Cystic Fibrosis, Part B
Enrollment: 32 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2017-12-18 (Actual); Study Completion 2017-12-18 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | 8 days
  To determine the incidence of treatment related adverse events.
Spirometry | 8 days
  To assess change from baseline spirometry.
Pulse Oximetry | 8 days
  To assess change in baseline pulse oximetry

SECONDARY OUTCOMES:
Observed maximum plasma concentration, taken directly from the individual concentration-time curve (Cmax) | Days 1, 2 and 8
  To characterize the pharmacokinetics of SNSP113
Area under concentration-time curve from time zero extrapolated to infinity (AUC) | Days 1, 2 and 8
  To characterize the pharmacokinetics of SNSP113

CONTACTS AND LOCATIONS:
Overall Officials: Maria Theresa Basco, MD, MPH, Study Director — Synspira, Inc.
Locations (2):
- United Kingdom (2):
  - Royal Brompton Hospital, London, England
  - Celerion, Belfast, Northern Ireland

IPD SHARING:
Plan to Share IPD: No